CLINICAL TRIAL: NCT07384767
Title: Efficacy and Safety of Topical Timolol in the Treatment of Cutaneous Surgical Wounds Left to Heal by Secondary Intention
Brief Title: Efficacy and Safety of Topical Timolol in Secondary Intention Surgical Wounds Healing
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2403423
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Mohs Micrographic Surgery; Excision Margin
Keywords: standard surgical excision; Mohs micrographic surgery; electrodesiccation and curettage; timolol; randomized
MeSH Terms: conditions — Margins of Excision | interventions — Timolol; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Timolol (Experimental): The treatment group will receive a topical timolol 0.5% solution, which will be applied to their wound daily for 12 weeks.
  Interventions: Drug: Timolol 0.5% Ophthalmic Solution
- Hydrogel (Placebo Comparator): The control group will receive standard care with the addition of hydrogel, which will also be applied to their wound daily for 12 weeks.
  Interventions: Other: Hydrogel of placebo

INTERVENTIONS:
Drug: Timolol 0.5% Ophthalmic Solution — Topical Timolol 0.5% solution will be applied to patients wounds in 2 cm intervals along the widest diameter of the wound daily for 12 weeks following their medical procedure.
  Arms: Timolol
Other: Hydrogel of placebo — Hydrogel will be placed on the wound at 2 cm intervals along the widest diameter of the wound daily for 12 weeks following the patient's medical procedure.
  Arms: Hydrogel

SUMMARY:
The purpose of this research study is to evaluate the efficacy and safety of topical timolol 0.5% for secondary intention wound healing following 1) Mohs micrographic surgery, 2) standard surgical excision, OR 3) electrodesiccation and curettage (ED&C). Please note that healing by secondary intention refers to when a wound heals naturally without surgical closure.

To evaluate the efficacy of topical timolol 0.5%, 220 participants will be recruited. Participants will be placed into one of two groups: The treatment group or the control group.

1. The treatment group will receive a topical timolol 0.5% solution, which will be applied to their wound daily for 12 weeks.
2. The control group will receive standard care with the addition of hydrogel, which will also be applied to their wound daily for 12 weeks.

During this 12-week period, both groups will be required to upload photos of their wound healing to their MyChart account at weeks 3, 6, 9, and 12. These photos will be reviewed by the investigator to assess wound healing. Re-epithelialization and earlier complete wound healing will be compared between both groups to determine the efficacy of topical timolol 0.5% solution compared to the standard of care.

DETAILED DESCRIPTION:
Secondary intention healing after cutaneous excisions or Mohs surgery is a commonly utilized technique in areas that are under high tension, in which primary closure would not be effective, or when patients defer a more complex closure technique. Secondary intention healing has drawbacks, as they take longer to heal and patients are left with a large wound at the surgical site for approximately 8 weeks. Topical timolol has shown promising results in lower extremity ulcers to improve wound healing, however larger trials on secondary intention surgical wounds have not been studied. This trial aims to fill this gap by comparing the efficacy and safety of topical timolol to standard wound care over a 12-week interval.

Participants who agree to the study, and who have opted to heal by secondary intention healing following their 1) Mohs micrographic surgery, 2) standard surgical excision, OR 3) electrodesiccation and curettage (ED&C) will be consented.

Once consented, the participant's demographics, medical history, and surgery details will be collected before being randomized into one of two groups: the treatment group or the control group.

1. The treatment group will receive a topical timolol 0.5% solution, which will be applied to their wound daily for 12 weeks.
2. The control group will receive standard care with the addition of hydrogel, which will also be applied to their wound daily for 12 weeks.

The participants and the research team will be blinded, meaning that they will not know which treatment the participant receives. Participants in both groups will be asked to upload photos of their wound healing at weeks 3, 6, 9, and 12 for the research team to examine.

The data will be analyzed to determine which group experienced faster re-epithelialization and earlier complete wound healing.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject of any race 18 years old or older
2. Patient opt to heal by secondary intention healing after discussion of reconstructive options following excision
3. Patients undergoing Mohs micrographic surgery, standard surgical excision, or electrodesiccation and curettage (ED&C) whose wounds are managed by secondary intention healing.
4. Willing to send photos of ulcer at 3 week intervals with ruler measuring length by width
5. Able to give informed consent themselves

Exclusion Criteria:

1. Cyst excisions (due to concern for inflammation)
2. Site shows evidence of infection (defined as a moderate or severe rating of all of the following clinical signs/symptoms: 1) increased warmth, 2) increased pain, 3) erythema, and 4) malodorous exudate at Screening or at Randomization (Visit 1), OR total organism count > 1 x 105 colony forming units (CFU) from the screening visit study ulcer culture sample)
3. Severe COPD/asthma/cardiac arrhythmia
4. Hx of documented beta blocker allergy
5. Cognitive impairment
6. Has medically documented history of Human Immunodeficiency Virus (HIV)
7. Has active malignancy on the study limb
8. Has immunodeficiency as defined by serum IgG, IgA, and IgM less than one-half the lower limit of normal
9. Has severe protein malnutrition as defined by serum albumin < 2.5 g/dL
10. Has serum aspartate aminotransferase (AST, SGOT, GOT) or serum alanine aminotransferase (ALT, SGPT, GPT) levels greater than twice the upper limit of normal
11. Has fatigue, palpitations, dyspnea, and/or angina at rest
12. Has a medically documented or self-reported history, within the previous 12 months from date of Screening Visit, of alcohol or drug abuse, particularly methadone or heroin
13. Has received previous treatment with the following during the 60 days prior to Screening: Immunosuppressive agents, radiation, chemotherapy, growth factors (epidermal growth factor, tumor necrosis factor, transforming growth factor, platelet derived growth factor, etc.)
14. Has received previous treatment with the following during the 30 days prior to screening: the site of the study ulcer, split- or full-thickness skin graft at the site of the study ulcer, biologically-active (or engineered) cellular or acellular product(s) at the site of the study ulcer, investigational drug or device
15. Has history of bradycardia (heart rate less than 60)
16. Has ESR>70mm/hr and CRP>100 mg/L at time of screening
17. Has medically documented history of hypotension/orthostatic hypotension and/or symptomatic hypotension (systolic blood pressure below 90 and diastolic blood pressure less than 60). (Note: There is no standard testing regimen protocol for orthostatic hypotension, even for patients starting on oral timolol)
18. Currently taking asthma or COPD medications (as documented in chart)
19. Has a medically documented diagnosis of myasthenia gravis, untreated hyperthyroidism, , Type 2, Type 3 heart block, cardiogenic shock, overt cardiac failure
20. Female who is pregnant or refuses to use adequate contraceptive methods and is of childbearing age during the trial
21. Prisoners, institutionalized individuals or vulnerable population

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Area of Surgical Ulcer | Baseline, week 3, week 6, week 9 and week 12
  The percent change in the area of surgical ulcers in patients using the study medication (treatment group) will be compared to those receiving standard care (placebo group).

SECONDARY OUTCOMES:
Infection Rate | Baseline to Week 12
  The number of patients who develop infections during treatment in both the treatment and placebo groups.
Risk Factor for Poor Wound Healing | Baseline to Week 12
  Sub-group analysis in patients with risk factors for poor wound healing; diabetes, smoking, cardiovascular disease, peripheral vascular disease, venous insufficiency, and/or long term prednisone use.
Type of Wounds | Baseline to Week 12
  Subgroup analyses will be performed by wound type (Mohs surgery, excision, ED&C) to assess for differential treatment effects.
Incidences of Hypotension | Baseline to Week 12
  Incidence of clinically significant hypotension (requiring medical attention) in patients treated with timolol
Incidences of COPD or Asthma Exacerbations | Baseline to Week 12
  Incidence of Chronic Obstructive Pulmonary Disease (COPD) or Asthma exacerbations in patients treated with timolol vs control.
Incidences of Hypertrophic Scar or Keloid | Baseline to Week 12
  The number of patients developing hypertrophic scar or keloid.
Incidences of Post Operative Bleeding | Baseline to Week 12
  The number of patients who developed post operative bleeding, and those who needed intervention by our clinic.
Use of Antibiotic | Baseline to Week 12
  The number of patients who started a topical or oral antibiotic during study treatment.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - VA Medical Center- Sacramento, Sacramento, California
  - UC Davis Health- Dermatology, Sacramento, California